CLINICAL TRIAL: NCT05589792
Title: The Effect of Acetazolamide on the Severity of REM Obstructive Sleep Apnea
Brief Title: Acetazolamide on REM OSA
Acronym: RemmOSA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ludovico Messineo, Instructor in medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022p002458
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule before bedtime for 3 nights before the studies (inclusive)
  Interventions: Drug: Placebo oral capsule
- Acetazolamide (Active Comparator): Acetazolamide 250 mg before bedtime 3 nights before the study, Acetazolamide 500 mg before bedtime for 2 nights before the study (inclusive)
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo before sleep for 3 nights before the study (inclusive)
  Arms: Placebo
Drug: Acetazolamide — Acetazolamide 250 mg 3 nights before the study at bedtime, Acetazolamide 500 mg for 2 nights before the study (inclusive) at bedtime.
  Arms: Acetazolamide

SUMMARY:
OSA is a highly prevalent disorder that has major consequences for cardiovascular health, neurocognitive function, risk of traffic accidents, daytime sleepiness and quality of life. In particular, REM sleep is accompanied by more frequent and longer obstructive events, that yield more profound hypoxemia than during non-REM (nREM). Exaggerated OSA severity in REM is the consequence of ventilatory drive dips, particularly during phasic eye movements. Unfortunately, the leading treatment for REM and nREM OSA, CPAP-which acts to pneumatically splint the pharynx open-is intolerable for many patients. Treatment outcomes for REM OSA are burdened by further incomplete CPAP adherence later in the night, which commonly leaves REM periods undertreated. In this protocol, the investigators will test the effect of Acetazolamide on REM OSA and on ventilatory parameters such as genioglossus muscle activity and ventilatory drive.

DETAILED DESCRIPTION:
After a baseline home sleep test that will assess the presence of OSA and REM OSA, two overnight, in-lab sleep studies will be performed: a drug night and a placebo night. The patient will breath spontaneously (without CPAP) for both nights. On the study nights, subjects will present to the laboratory in the evening and be instrumented with a full polysomnigraphy for monitoring sleep, physiological variables (endotypes), and respiratory events. Participants will also be instrumented with EMG wires and introesophageal catheter for the recording of genioglossus muscle activity and respiratory drive, respectively. A history and physical examination will be performed on each night prior to beginning the study, as will a urine pregnancy test in premenopausal women. Acetazolamide 500 mg will be taken for 2 days (including the day of the study), after a day in which it will be administered at half dose, before bedtime. Subjects will sleep at least 50% of the night in the supine position. At least four hours of sleep with high quality signal acquisition will be required for a study to be judged adequate. Subjective sleep quality will be assessed in the morning. After the first overnight study is completed, there will be a four day washout period prior to crossing over to the other treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed REM OSA (per baseline screening: REM AHI/nREM AHI≥2) [31-33]
* REM duration>10 minutes
* Not using CPAP (>1 week).

Exclusion Criteria:

* Any uncontrolled medical condition
* Current use of the medications under investigation
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Conditions likely to affect obstructive sleep apnea physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Respiratory disorders other than sleep disordered breathing:

chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.

* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Contraindications for acetazolamide, including:

  * Hyperchloremic acidosis
  * Hypokalemia
  * Hyponatremia
  * Adrenal insufficiency
  * Impaired kidney function
  * Hypersensitivity to acetazolamide or other sulfonamides.
  * Marked liver disease or impairment of liver function, including cirrhosis.
* Contraindications to the use of lidocaine 4%/oxymetazoline HCT.
* Claustrophobia
* Pregnancy or nursing

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | 1 night
  Number of events/hour of sleep
Hypoxic burden | 1 night
  The total area under the respiratory event-related desaturation curve, measured as in %min/hr
Ventilatory drive in REM and NREM | 1 night
  Ventilatory drive will be calculated using diaphragm EMG (as percent of eupneic ventilatory drive)
Genioglossus activity in REM and NREM | 1 night
  Genioglossus activity will be calculated using EMG wires under the tongue (as percent of eupneic activity or maximal activity)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No